CLINICAL TRIAL: NCT06967545
Title: A One-Arm Open Trial of a Smartphone Delivered Treatment for Suicidal Thoughts and Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Adam C. Jaroszewski, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P003049-phase1
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Suicide Attempt; Suicide Ideation
Keywords: Suicide; Ecological momentary assessment (EMA); Therapeutic Evaluative Conditioning (TEC)
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smartphone-delivered active Therapeutic Evaluative Conditioning for Suicide (active TEC) (Experimental): Optional smartphone-delivered active Therapeutic Evaluative Conditioning for Suicide (active TEC-S) for 30 days.
  Interventions: Behavioral: Smartphone-delivered Therapeutic Evaluative Conditioning for Suicide (TEC-S)

INTERVENTIONS:
Behavioral: Smartphone-delivered Therapeutic Evaluative Conditioning for Suicide (TEC-S) — Therapeutic Evaluative Conditioning for Suicide (active TEC-S) is a behavioral treatment where participants are given optional access to a computerized task/game where they repeatedly pair suicidal behavior stimuli (pictures, words) with other negative stimuli and self-related stimuli with positive stimuli.

SUMMARY:
This study aims to evaluate the acceptability, safety, and preliminary efficacy of a smartphone-delivered intervention called Therapeutic Evaluative Conditioning for Suicide (TEC-S) in reducing suicidal thoughts and behaviors (STB) among adults with recent and frequent suicide ideation.

DETAILED DESCRIPTION:
The present study is a one-arm open trial designed to evaluate the safety, acceptability, and preliminary efficacy of Therapeutic Evaluative Conditioning for Suicide (TEC-S), a smartphone-delivered intervention aimed at reducing suicidal thoughts and behaviors (STB). Participants in this study will be 20 adult participants (ages 18+) who report recent and frequent STB, residing within the greater-Boston, MA area.

Participants will receive 3x/daily EMA and optional access to active TEC-S. Evaluative conditioning uses classical conditioning to alter attitudes. The aim of TEC-S is to alter attitudes toward suicide and, in turn, reduce STB. EMAs will monitor STB, safety, and acceptability, and efficacy. Weekly behavioral and self-report assays will assess hypothesized treatment mechanisms. The study's aim is to evaluate the safety, acceptability, and preliminary efficacy of Therapeutic Evaluative Conditioning for Suicide (TEC-S).

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18+
* Relatively frequent and recent (≥5 days within the past-month) active suicidal thoughts as assessed via SITBI-R.
* Willing and able to provide at least one emergency contact (name, phone number, relation).
* Owns an Android or iOS smartphone.
* Possesses at least occasional access to Wi-Fi-enabled internet for data down/uploads.
* Fluent in English and willing to provide informed consent.
* Living in the Boston metropolitan area (i.e., ~50 mile radius around Boston, MA)

Exclusion Criteria:

* Recent (past 3-month) hypo/manic symptoms or homicidal ideation or lifetime psychosis spectrum diagnosis as assessed via MINI 7.0.2.
* Recent acute suicide risk operationalized as affirmative responses to BOTH below items during structured clinical interview AND evaluation by the PI in consultation with Mentors/Advisor Drs. Wilhelm, Kleiman, and/or Bentley:
* At any time in past week: ≥ 8/10 current intent to act on suicidal thoughts (0 ["not at all"] to 10 ["extremely strong"]); AND
* At any time in past week: thought of a specific suicide plan (i.e, known method/means and/or location) with access to lethal means
* Impaired vision (e.g., legal blindness), technological illiteracy, or intellectual disability that might impair ability to provide valid data and/or informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
TEC-S Acceptability | Through completion of treatment phase (day 1 through 30)
  (i) Indexed as the proportion of TEC-S sessions accessed within the first week, (ii) adapted items from the Credibility/Expectancy Questionnaire (CEQ), rated on a 9-point scale. : "How satisfied were you with your overall experience with TEC-S?" "How satisfied were you with your understanding of how to complete TEC-S (iii)End-User Mobile Application Rating Scale (uMARS), with items rated on a 5-point scale.
TEC-S Safety | Through completion of treatment phase (day 1 through 30)
  Changes in suicide-related thoughts (e.g., intent, desire, urge, preparation) and affective responses (e.g. stress) before and after randomized stimuli in each TEC-S session, assessed via ecological momentary assessment

SECONDARY OUTCOMES:
Desire to die by suicide (Likert) | Through completion of treatment phase (day 1 through 30)
  Right now, how strongly do you want to kill yourself? [0 (not at all) to 10 (extremely)
Suicide urge (Likert) | Through completion of treatment phase (day 1 through 30)
  Right now, how strong is your urge to kill yourself [0 (not at all) to 10 (very strong)]; assessed via 3x/day ecological momentary assessment.
Suicide thought incidence | Through completion of treatment phase (day 1 through 30)
  Since the last survey, have you had suicidal thoughts? (yes/no); assessed daily via ecological momentary assessment
Suicide preparation incidence | Through completion of treatment phase (day 1 through 30)
  Since the last survey, have you made any preparations to kill yourself? (yes/no); assessed daily via ecological momentary assessment.
Suicide attempt incidence | Through completion of treatment phase (day 1 through 30)
  Since the last survey, have you attempted to kill yourself? (yes/no); assessed daily via ecological momentary assessment
Suicidal behaviors (composite) | Through completion of treatment phase (day 1 through 30)
  A composite variable consisting of (i) suicide plan incidence, (ii) suicide preparation incidence, (iii) suicide attempt incidence, each assessed via ecological momentary assessment
Suicidal aversion (AMP) | Through completion of treatment phase (day 1 through 30)
  Suicide aversion assessed implicitly/behaviorally via the Affect Misattribution Procedure (AMP)
Suicidal aversion (Likert) | Through completion of treatment phase (day 1 through 30)
  Valence ratings of suicide-related pictures using a 9-point scale (-4 [extremely unpleasant] to 0 [neutral] to 4 [extremely pleasant]); assessed weekly.
Suicidal affection (AMP) | Through completion of treatment phase (day 1 through 30)
  Self affection assessed implicitly/behaviorally via the Affect Misattribution Procedure (AMP)
Suicide intent (Likert) | Through completion of treatment phase (day 1 through 30)
  Right now, how strong is your intention to kill yourself today? [0 (I am definitely not going to kill myself today) to 10 (I am definitely going to kill myself today)]; assessed via 3x/day ecological momentary assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States